CLINICAL TRIAL: NCT06188897
Title: Biomechanical Relationship Between Trunk Flexion and Mouth Opening: Pilot Study
Acronym: REFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Laura Menés Fernández, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23/2016
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Hamstring Injury; Temporomandibular Joint Disorders; Stretch
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group did the intervention, which consisted of self-stretching of the masticatory muscles. This stretch consisted of introducing three knuckles of the non-dominant hand between the incisors for two minutes while sitting
  Interventions: Other: Self-stretching of the masticatory musculature
- Control group (Placebo Comparator): The control group was asked to introduce only two knuckles in the oral cavity and perform a mandibular occlusion, an intervention that serves as a simulated stretch in said group.
  Interventions: Other: Control group intervention

INTERVENTIONS:
Other: Self-stretching of the masticatory musculature — If the subject belonged to the Treatment group, he was instructed to self-stretch the masticatory muscle.
  This stretch consisted of introducing three knuckles of the non-dominant hand between the incisors for two minutes while sitting.
  Arms: Experimental group
Other: Control group intervention — The control group was asked to introduce only two knuckles in the oral cavity and perform a mandibular occlusion, an intervention that serves as a simulated stretch in said group.
  Arms: Control group

SUMMARY:
The aim of the present study is to analyze if there is a biomechanical relationship between trunk flexion and buccal opening and to observe if there is an improvement of trunk flexion by performing the "sit and reach" test when stretching the masticatory muscles.

DETAILED DESCRIPTION:
The study design is made up of a double-blind clinical trial with 60 participants randomly divided into two groups of 30 people each (Treatment group and Control group). Basal measurements of the mouth opening were taken with a vernier caliper and the trunk flexion measurements were taken by means of the "sit and reach" test. These measurements were carried out again after the intervention, which consisted of self-stretching of the masticatory muscles for the Treatment group and an occlusion of the mouth for the Control group. In the results there was an increase in the trunk flexion compared to the initial values in both groups (Treatment group 2.8 (1.51), Control group 1.97 (2.31) and this increase was greater in the Treatment group even though the difference with the Control group was not statistically significant. Therefore, the stretching of the masticatory muscles does not cause an immediate increase in the degree of trunk flexion measured by the "sit and reach" test. As a consequence, we cannot confirm the existence of a biomechanical relationship between trunk flexion and mouth opening.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18 and 26 years old (both included).
2. Having signed the consent form.
3. Being able to introduce three knuckles of the non-dominant hand between the incisors.

Exclusion Criteria:

1. Having a musculoskeletal injury in the lower extremity and / or in the jaw.
2. Being in the process of receiving physiotherapy treatment and / or having undergone any odontologic or maxillofacial surgery in the last month.
3. Having suffered dislocations, painful clicks or being diagnosed with some type of temporomandibular joint (TMJ) dysfunction.
4. Having hypermobility in the temporomandibular joint (TMJ) that is, the measurement of the buccal opening being greater than 60 mm.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Trunk flexion | 1 year
  Trunk flexion in cm, taken by using the "sit and reach" drawer (Eve-que). The measurements were made three consecutive times with an interval of five seconds between them. The result of the arithmetic average of the three measurements was the one that was accounted for in the study. For the measurement of trunk flexion, the subject was placed on the floor with his back against the wall and having the soles of both feet in contact with the drawer.

SECONDARY OUTCOMES:
Mandibular opening | 1 year
  Mandibular opening in mm., assessed using the vernier caliper (INCUTEX Germany GmbHl). The measurement was made three consecutive times with an interval of five seconds between them. The result of the arithmetic average of the three measurements was the one that was caliper (corresponding to 0 of the ruler) was placed at the upper end of the lower central incisors and measured to the edge of the corresponding central incisor.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Menés Fernández, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espejo-Antunez L, Castro-Valenzuela E, Ribeiro F, Albornoz-Cabello M, Silva A, Rodriguez-Mansilla J. Immediate effects of hamstring stretching alone or combined with ischemic compression of the masseter muscle on hamstrings extensibility, active mouth opening and pain in athletes with temporomandibular dysfunction. J Bodyw Mov Ther. 2016 Jul;20(3):579-87. doi: 10.1016/j.jbmt.2015.12.012. Epub 2016 Jan 7. PMID 27634081
- [Background] Rodriguez-Blanco C, Cocera-Morata FM, Heredia-Rizo AM, Ricard F, Almazan-Campos G, Oliva-Pascual-Vaca A. Immediate Effects of Combining Local Techniques in the Craniomandibular Area and Hamstring Muscle Stretching in Subjects with Temporomandibular Disorders: A Randomized Controlled Study. J Altern Complement Med. 2015 Aug;21(8):451-9. doi: 10.1089/acm.2014.0332. Epub 2015 Jun 2. PMID 26218883